CLINICAL TRIAL: NCT02557659
Title: Clinical Investigation Plan for the Zenith® Low Profile AAA Endovascular Graft
Brief Title: Zenith® Low Profile AAA Endovascular Graft
Status: No longer available | Type: Expanded Access
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 08-013 CA
Record Dates: First submitted 2015-09-22; First posted 2015-09-23 (Estimated); Last update posted 2018-03-12 (Actual); Status verified 2018-03

CONDITIONS: Abdominal Aortic Aneurysms; Iliac Aneurysms; Aorto-iliac Aneurysms
Keywords: Low Profile; Abdominal Aortic Aneurysms; Endovascular
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Iliac Aneurysm

INTERVENTIONS:
Device: Zenith Low Profile AAA Endovascular Graft — Treatment of patients with abdominal aortic, aorto-iliac, or iliac aneurysms having morphology suitable for endovascular repair

SUMMARY:
This extended investigation is to provide continued physician access to the device and collect confirmatory safety and effectiveness data.

ELIGIBILITY:
Inclusion Criteria:

•Subject has at least one of the following

* Aortic or aortoiliac aneurysm
* Iliac aneurysm
* Aneurysm with a history of growth

Exclusion Criteria:

* Less than 18 years of age
* Inability or refusal to give informed consent
* Life expectancy less than 2 years
* Pregnant of breastfeeding or planning on becoming pregnant with 60 months
* Unwilling to comply with the follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Fairman, MD, Principal Investigator — University of Pennsylvania
Locations (22):
- United States (22):
  - University of California San Francisco-VA, San Francisco, California
  - University of California, San Francisco, San Francisco, California
  - Stanford University Medical School, Stanford, California
  - Yale New Haven School of Medicine, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Massachusetss General Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Morristown Memorial Hospital, Morristown, New Jersey
  - New York University - Langone Medical Center, New York, New York
  - New York Presbyterian Hospital - Cornell, New York, New York
  - New York Presbyterian - Columbia, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio Health Research Institute, Columbus, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Washington-Harborview Medical Center, Seattle, Washington
  - Aurora Saint Luke's Medical Center, Milwaukee, Wisconsin